CLINICAL TRIAL: NCT05931679
Title: Pandemic-Proofing Simulation-based Education: Development and Evaluation of Interactive Virtual Educational Content for Medical Trainees
Brief Title: Pandemic-Proofing Simulation-based Education
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Sunnybrook Research Institute (Other)
Responsible Party: Principal Investigator, Glenn Posner, Associate Professor, Division of General Obstetrics and Gynecology, Ottawa Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 20210197-01H
Record Dates: First submitted 2022-05-11; First posted 2023-07-05 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: COVID 19
Keywords: Virtual Reality; Simulation
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of three groups - interactive VR, 360o video, or theatre-based education.
Who Masked: Participant
Masking Description: Participant will receive a unique study ID which will be used throughout the life of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Interactive VR (Active Comparator): a virtual classroom - learners wearing VR headsets in the safety of their home are immersed in a computer-generated simulation centre. Through their avatars, they can interact from a first-person perspective with their environment, colleagues and instructors. The virtual patient has been in a car accident and the learners, by interacting with the virtual trauma bay environment, must work together to perform a primary trauma survey and resuscitate the patient. The interactive VR environment provides the team with real time information (e.g. oxygen saturation levels, heart rate) in a realistic environment that includes the uncertainty, noise, and time pressures of a real case.
  Interventions: Device: VR Headset
- 360 degree video (Active Comparator): An immersive environment based on high-definition 360o video obtained from our simulation centre. Single learners, wearing a VR headset, find themselves in the resuscitation room, at the foot of the bed, leading a trauma team through the assessment and resuscitation of a patient in a virtual choose-your-own-adventure scenario. At several key points in the videos, learners are presented with interactive decision points, and their choices determine how the rest of the video unfolds.
  Interventions: Device: VR Headset
- Theatre-based education (Active Comparator): Traditional theatre-based simulation sessions require the physical presence of interdisciplinary groups of learners caring for a physical mannequin-based patient, where social distancing is challenging.
  Interventions: Other: Traditional Theatre-based simulation

INTERVENTIONS:
Device: VR Headset — A VR headset will be used for participants in the Interactive VR and 360 degree video groups.
  Arms: 360 degree video; Interactive VR
Other: Traditional Theatre-based simulation — Traditional theatre-based simulation sessions require the physical presence of interdisciplinary groups of learners caring for a physical mannequin-based patient, where social distancing is challenging.
  Arms: Theatre-based education

SUMMARY:
The goal is to develop and evaluate two VR simulations (interactive VR, 3600 video) applied to the context of Emergency Medicine. The aim of this pilot study is to develop two VR simulations, and to compare their effectiveness with traditional theatre-based simulations.

Primary Objectives: to compare knowledge retention and application of knowledge during emergency crisis scenarios following VR-360, interactive VR and theatre-based simulation sessions.

Secondary Objectives: to assess the usability and feasibility (resources), as well as the emotional engagement, of the above three modalities.

DETAILED DESCRIPTION:
Phase 1: Creation of Content: A software engineer with expertise in video-game development will be hired to develop the computer-generated emergency department in collaboration with the educators and clinicians on the team. A theatre-based trauma scenario from the current uOttawa Emergency Department curriculum will be adapted to the VR platform. This virtual environment will allow a team of students to manage a patient simultaneously through their avatars, from a first-person perspective. In parallel, the same scenario will be scripted, in all its permutations, and recorded using a 360-degree HD video camera. The recording will be made using the investigators as actors, with additional interprofessional volunteers recruited as needed. These videos will be edited and then converted to an application that can be uploaded to the Oculus platform. Both platforms will undergo piloting for content and usability. The amount of time, money and other resources required to develop each of these scenarios will be calculated.

Phase 2: Evaluating the intervention:

Pre-test: Prior to participating in one of the 3 educational interventions, participants will complete a pre-test of their content-specific knowledge and knowledge application with respect to trauma resuscitation. As well, they will participate in a video-recorded in-situ simulation of a trauma resuscitation. Team performance will be recorded for subsequent scoring (see measures and analysis section below). During the in-situ sessions, the investigators will measure the learners' heart rate (HR) and heart rate variability (HRV) with the use of a Polar H10 chest belt linked with a commercial capture and analysis software program on an iPad. This will allow us to measure both arousal and stress responses, as physiological indication of the learners' emotional engagement.

Intervention: Following the pre-test, residents will either participate in the interactive VR, the 360o video or the in-person theatre-based simulation sessions.

Post-test. Two weeks after the education session, all participants will complete a post-test of their knowledge and knowledge application (matched in difficulty with pre-test), as well as lead an in-situ simulated trauma resuscitation. The sessions will be videotaped for subsequent rating of clinical and team performance.

ELIGIBILITY:
Inclusion Criteria:

Participants will be residents or medical students

Exclusion Criteria:

Anyone who is not a resident or medical student

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measures will be changes in knowledge and in clinical performance from pre-test to post-test. | Two weeks, will be done prior to post-test of knowledge and Knowledge application
  Two experienced trauma resuscitation instructors will view and score the videos independently, blinded to the group allocation and whether the scenario is pre or post the intervention. The raters will evaluate the learners using the Ottawa Global Rating Scale which is a 7 point anchored ordinal scale for performance in five major categories of Crisis Resource Management (CRM) and an overall performance. The score provides 12 items in five category of CRM with a maximum score of 30 points. The higher the number of points, the "better" the individual's performance (better outcome).

SECONDARY OUTCOMES:
Mean heart rate (HR) | During the simulation sessions, throughout the study: 5 minutes prior to start of each scenario, for the duration of each scenario, for the duration of the debriefing, for the duration of the post-test over a 2 week period
  The investigators will compare arousal levels between the 3 experimental conditions (interactive VR, 360o video, theatre-based) by heart rate monitoring. Continuous heart rate (R-R intervals) will be measured with the POLAR® H10 device, a non-invasive chest strap with a transducer worn directly against the sternum paired with a smart device application (EliteHRV). The participants heart rate will be recorded for 5 minutes prior to start of each scenario (Pre-scenario - to capture anticipatory stress responses), for the duration of the debriefing (divided into sequential 5 min periods), for the duration of the post-test (divided into sequential 5 min periods]. For each participant, the investigators will analyse the participant's mean heart rate (averaged over each measured time period)..
Peak heart rate (HR) | During the simulation sessions, throughout the study: 5 minutes prior to start of each scenario, for the duration of each scenario, for the duration of the debriefing, for the duration of the post-test over a 2 week period
  The investigators will compare arousal levels between the 3 experimental conditions (interactive VR, 360o video, theatre-based) by heart rate monitoring. Continuous heart rate (R-R intervals) will be measured with the POLAR® H10 device, a non-invasive chest strap with a transducer worn directly against the sternum paired with a smart device application (EliteHRV). The participants heart rate will be recorded for 5 minutes prior to start of each scenario (Pre-scenario - to capture anticipatory stress responses), for the duration of the debriefing, for the duration of the post-test. For each participant, the investigators will analyse the participant's peak heart rate over each time period.
Heart rate variability - rMSSD | During the simulation sessions, throughout the study: 5 minutes prior to start of each scenario, for the duration of each scenario, for the duration of the debriefing, for the duration of the post-test
  The investigators will compare individual stress scores between the 3 experimental conditions (interactive VR, 360o video, theatre-based) by heart rate variability (HRV) monitoring. Continuous heart rate (R-R intervals) will be measured with the POLAR® H10 device, a non-invasive chest strap with a transducer worn directly against the sternum paired with a smart device application (EliteHRV). The participants HRV will be recorded for 5 minutes prior to start of each scenario (Pre-scenario - to capture anticipatory stress responses), for the duration of the debriefing (divided into sequential 5 min periods), for the duration of the post-test (divided into sequential 5 min periods]. For each participant, the investigators will analyse the participant's root mean square of successive R-R interval differences (rMSSD).
Heart rate variability - pNN50 | During the simulation sessions, throughout the study: 5 minutes prior to start of each scenario, for the duration of each scenario, for the duration of the debriefing, for the duration of the post-test over a 2 week period
  The investigators will compare individual stress scores between the 3 experimental conditions (interactive VR, 360o video, theatre-based) by heart rate variability (HRV) monitoring. Continuous heart rate (R-R intervals) will be measured with the POLAR® H10 device, a non-invasive chest strap with a transducer worn directly against the sternum paired with a smart device application (EliteHRV). The participants HRV will be recorded for 5 minutes prior to start of each scenario (Pre-scenario - to capture anticipatory stress responses), for the duration of the debriefing (divided into sequential 5 min periods), for the duration of the post-test (divided into sequential 5 min periods]. For each participant, the investigators will analyse the participant's percentage of successive R-R intervals that differ by more than 50Ms (pNN50).

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Posner, Principal Investigator — Ottawa Hospital Research Institute

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2023-04-15): https://cdn.clinicaltrials.gov/large-docs/79/NCT05931679/Prot_000.pdf
  • Informed Consent Form (2021-10-27): https://cdn.clinicaltrials.gov/large-docs/79/NCT05931679/ICF_001.pdf